CLINICAL TRIAL: NCT04292184
Title: Evaluation of Thiosulfate in End Stage Renal Disease and Kidney Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Alp Sener, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 112145
Record Dates: First submitted 2019-05-23; First posted 2020-03-03 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: End Stage Renal Disease (ESRD)
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — sodium thiosulfate

STUDY DESIGN:
Intervention Model Description: For the purposes of this study we will flush the deceased donor kidney with UW (perfusion solution) or UW + sodium thiosulfate (STS). There will be two groups in the study - UW with or without STS and patients will be randomly assigned to a group in a 1:1 ratio (i.e. 50 in one group and 50 in the other).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UW (perfusion solution) + sodium thiosulfate (STS) (Active Comparator): We will flush the deceased donor kidney with UW (perfusion solution) + sodium thiosulfate (STS)
  Interventions: Drug: Seacalphyx (sodium thiosulfate pentahydrate injection BP) 25%
- UW (perfusion solution) (No Intervention): Kidney will be flushed with UW (perfusion solution) which is the normal standard of care.

INTERVENTIONS:
Drug: Seacalphyx (sodium thiosulfate pentahydrate injection BP) 25% — The kidney will have 100 mL of 500µM STS added directly to the existing pulsatile perfusion solution at 4°C.
  Other Names: Sodium thiosulfate (STS)
  Arms: UW (perfusion solution) + sodium thiosulfate (STS)

SUMMARY:
Kidneys retrieved from deceased donors will be randomized for conventional perfusion (University of Wisconsin: UW) with or without supplementation of thiosulfate, a major H2S metabolite, and transpl anted thereafter. Recipient's renal function will be assessed prospectively to determine if thiosulfate improves allograft function.

DETAILED DESCRIPTION:
The rise in the incidence of end stage renal disease (ESRD) is both a national and international concern. Renal transplantation is currently the best available treatment for established renal failure as it not only offers freedom from dialysis but improves survival, provides better quality of life and is more cost effective.1 Unfortunately there is a widening discrepancy between the incidence of ESRD and the number of available organs for transplantation. The number of organs available from these donors has never been sufficient for all of the patients on the transplant waiting lists. Over the past decade, donation after cardiac death (DCD) has gained popularity as a method to increase the number of organs available for transplantation. As expected, our attempts at maximizing usable organs for transplant with DCD kidneys comes at a price with a higher risk of delayed graft function (DGF) and graft loss compared to kidneys from standard criteria donors.2 Given that the DCD group is inherently plagued by longer warm ischemic times and labile cardiovascular physiology at the time of the donor operation, up to 30% of recipients of DCD kidneys lose their renal grafts within 5 years and up to 50% in 10 years.3,4 This results in up to 25% of those patients going back onto renal replacement therapies and then becoming relisted for transplantation. If current trends continue, the deficit in organ allocation is expected to rise over the next 20 years due to projected global incidences of obesity, diabetes and hypertension5, which will lead to an increased use of organs procured from increasingly marginal donors to keep up with the demand.

Ischemia reperfusion injury (IRI) is a complex biological process involving cell death, microcirculatory compromise, altered transcription, inflammation and immune activation. Modulation of IRI particularly in DCD organs (characterized by prolonged warm ischemia followed by periods of long hypothermic storage), could impact both short and long term patient and graft outcomes. Importantly, IRI affects all donor kidneys, but the effect appears to be greatest in the DCD cohort. Indeed, significant efforts have been applied in the experimental and pre-clinical setting to develop strategies to ameliorate the negative effects of IRI.

However, there is currently no active pharmacological agent used during transplantation to reduce the impact of IRI. Efforts to curb IRI during transplantation have involved either pulsatile (machine perfusion) or static storage of donor kidneys in various preservation solutions at hypothermic (4ºC) conditions during the peri-transplant period. Hypothermia slows cellular metabolism and subsequent ATP depletion during the ischemic period, while organ preservation solutions contain a myriad of electrolytes and other solutes which help to maintain osmotic conditions, scavenge free radicals and stimulate cellular metabolism upon reperfusion. University of Wisconsin (UW) solution is the most commonly used preservation solutions that has been shown to be the most effective at decreasing the risk of DGF following renal transplantation.6 H2S has long been known for its unsavory "rotten eggs" smell and toxic effects at high concentrations. However, it has been later discovered that H2S is also produced endogenously in mammalian cells mainly via the metabolism of L-cysteine by two cytosolic enzymes, cystathionine ß-synthase (CBS) and cystathionine -lyase (CSE) and one mitochondrial enzyme, 3-mercaptopyruvate sulfurtransferase (3-MST).

Various H2S donation strategies have been developed and tested in vitro and in vivo. The two most often used salts NaHS and Na2S, are among the simplest sources of H2S. They dissociate very rapidly at physiological pH to generate H2S. The resulting bolus of instantly generated H2S does not mimic the endogenous, constitutive enzymatic synthesis of small amounts of H2S.7-9 Another possibility is the use of sodium thiosulphate (Na2S2O3, STS), a major metabolite of H2S, commercially available compound and typically available as the pentahydrate, Na2S2O3·5H2O. It also has functions as a preservative in table salt (less than 0.1 %) and alcoholic beverages (less than 0.0005 %). While these amounts are very small, they indicate that the general population is consuming STS (Sodium thiosulfate) on a regular basis and increasing the dose may have important therapeutic applications, especially in ESRD and chronic kidney disease patients.

In clinical studies, STS has been used in the treatment of some rare medical conditions including calciphylaxis in hemodialysis patients with end-stage kidney disease10,11. Moreover, short term therapeutic use of STS has been proven safe12. STS is also proposed to be an antioxidant10 and HC-approved for use in cyanide poisoning13,14or cisplatin toxicity15. Furthermore, vasodilating properties of STS itself have been described16. However, the effect of STS on the protection of kidney injury and renal graft function post transplantation has not been described clearly. We hypothesize that supplementation of preservation solutions with STS will inhibit IRI injury, improve renal function and graft survival in kidney transplant recipients and that this effect will be heightened in recipients receiving kidneys obtained from DCD donors.

ELIGIBILITY:
Inclusion Criteria:

- All patients >18years old who are being considered for renal transplantation at LHSC that are receiving a DCD kidney.

Exclusion Criteria:

* Age <18 years old
* Inability to give informed consent,
* Patients receiving kidneys from living donors
* Patients with known hypersensitivity to either SEACALPHYX or to any of the ingredients contained within.
* Pregnant women.
* Patients with sulfite allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-03-21 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Patient urine output | 1 week
  1 week following transplant
Change in Patient urine output | 1 year
  between 1 week and 1 year following transplant
Serum Creatinine | 1 week after transplant
  Patient Blood serum creatinine results
Slow Graft Function | 1 week after transplant
  Patients' Rate of slow graft function
eGFR | 1 week after transplant
  Patient eGFR Results

SECONDARY OUTCOMES:
Biopsy proven Acute tubular necrosis (ATN) | 1 week
  Measuring death of tubular epithelial cells that form the renal tubules of the kidneys.
Urine protein/creatinine ratio | 1 week
  Patient Urine protein/creatinine ratio results
Urinary injury biomarkers (KIM-1/NGAL). | 1 week
  Patient urinary injury biomarkers (KIM-1/NGAL).

CONTACTS AND LOCATIONS:
Overall Officials: Alp Sener, Dr., Principal Investigator — LHSC
Locations (1):
- London Health Sciences Centre, University Hospital, London, Ontario, Canada